CLINICAL TRIAL: NCT03577925
Title: The Standard Mangagement of High-Risk HPV Infection During Follow-up Visits
Brief Title: The Standard Management of HPV Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Yu mei Wu, Yu mei Wu, Capital Medical University
Other Study IDs: ZYLX201705
Record Dates: First submitted 2018-06-24; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: the High-Risk HPV Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HSIL: the patients with HSIL
  Interventions: Diagnostic Test: HPV genotype test
- stage IA1 cervical squamous cancer: the patients with stage IA1 cervical squamous cancer
  Interventions: Diagnostic Test: HPV genotype test

INTERVENTIONS:
Diagnostic Test: HPV genotype test — HPV genotype test is a diagnostic test by smearing the cervix to find out whether a patient is hpv infected, and if infected, the test can descover the concrete hpv genotype.

SUMMARY:
High-risk human papillomavirus (HR-HPV) infection is a necessary condition in the occurence and development of cervical squamous intraepithelial lesion (SIL) and cervical cancer. There are cases that high-grade SIL (HSIL) and stage IA1 cervical squamous cancer remain or reoccur, or even become more severe after conization. The infection situation of HR-HPV, which plays an important role in the prognosis of cervical lesion, should be consulted in the management and follw-up after conization. It is worthwhile making further study in the specific practical significance of the HR-HPV in the prognosis of cervical lesion, as well as the high-risk factors that influence the prognosis of HR-HPV.

DETAILED DESCRIPTION:
Main purpose:To work out the standard management of HPV infection by following up the HPV infection situation of the patients with high-grade SIL (HSIL) and stage IA1 cervical squamous cancer after conization.

Research design:First, to do the retrospective analysis toward the patients who received conization between Jan 2009 to Aug 2016.Second,to do the prospective analysis toward the patients who received conization between Spt 2016 to Aug 2018.

Inclusive criteria of study population:The patients who had finished HPV genotype testing before conization;who had never received treatment other than conization;who were histologically diagnosed as HSIL or IA1 cervical squamous cancer;who had not been diagnosed as any cervical diseases before;who were under age 70;who did not have any severe diseases that influence the follow-up.

Follow-up methods:to do the follow-up to the target patients by 3,6,9,12,18,24 months after conization.

Follow-up contents:the HR-HPV genotype infection before conization;the grade of lesion;the age when received conization;the gravity and parity;the situation of the glands invovement

ELIGIBILITY:
Inclusion Criteria:

* age not above 70
* histologically diagnosed as HSIL or stage IA1 cervical squamous cancer
* received conization in Beijing Obstetrics and Gynecology Hospital
* HR-HPV infected without any treatment other than conization
* HR-HPV genotype tested before coniztion

Exclusion Criteria:

* age above 70
* with severe desease that influence the follow-up
* received other treatment on cervical lesion
* data incompleted
* not meet the inclusive criteria

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the HR-HPV genotype tested positive patients with HSIL or stage IA1 cervical squamous cancer who received conization at genocology oncology department in Beijing Obstetrics and Gynecology Hospital during Oct 2016 to Oct 2018.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
The HR-HPV clearance | 24 months
  The difference of the HR-HPV clearance between HSIL and stage IA1 cervical squamous cancer

CONTACTS AND LOCATIONS:
Overall Officials: Yu mei Wu, Doctor, Study Director — Beijing Obstetrics and Gynecology Hospital
Locations (1):
- Yu mei Wu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided